CLINICAL TRIAL: NCT00914654
Title: Blood and Urinary Concentrations of Inhaled Formoterol in Asthmatic Subjects and Elite Athletes With Asthma
Brief Title: Concentrations of Formoterol in Blood and Urine
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bispebjerg Hospital (Other)
Collaborators: Hormone Laboratory, Aker University Hospital, Oslo, Norway (Other)
Responsible Party: Jimmi Elers, Bispebjerg Hospital, Respiratory Research Unit
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: FOR2009JE; EudraCT number 2009-012039-14
Record Dates: First submitted 2009-06-04; First posted 2009-06-05 (Estimated); Last update posted 2009-06-05 (Estimated); Status verified 2009-06

CONDITIONS: Asthma
Keywords: Asthma; Doping; Formoterol; Urinary concentrations; Beta-agonists
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Healthty (Other): 10 healthy men
  Interventions: Drug: inhaled formoterol
- Asthmatics (Other): 10 male asthmatic subjects
  Interventions: Drug: inhaled formoterol
- Elite asthmatics (Other): 10 male elite athletes with asthma
  Interventions: Drug: inhaled formoterol

INTERVENTIONS:
Drug: inhaled formoterol — Inhalation of 18 microgram formoterol as one dose. Oxis Turbohaler 9 microg/dose, MA no. 30072.
  Other Names: Oxis Turbohaler 9 microg/dose, MA no. 30072.

SUMMARY:
The purpose of the study is to assess the blood and urine concentrations of inhaled formoterol.

DETAILED DESCRIPTION:
The purpose of the study is to assess the serum and urine concentrations after inhalation of 18 microgram formoterol as one dose.

Furthermore to investigate the serum and urine concentrations of inhaled formoterol and evaluate the difference between three groups: healthy men, male asthmatic subjects and male elite athletes with asthma.

ELIGIBILITY:
Inclusion Criteria:

* Physician-diagnosed asthma with positive reversibility or challenge test.
* Informed consent.
* Age between 18-45 years.
* Sex: male.
* Asthma classified as mild to moderate according to GINA guidelines.
* Used beta-2-agonist in minimum 12 months.

Exclusion Criteria:

* Smokers or ex-smokers with a smoking history of 10 pack years or more.
* Respiratory tract infections within the last 2 weeks prior to study day.
* Subjects with other chronic diseases than asthma and allergy.
* Allergy towards the study medicine.
* Use of beta-2-agonist 10 days prior to study day.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-07; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Serum and urine concentrations of formoterol | baseline, 4, 8, and 12 hours after medicine administration

CONTACTS AND LOCATIONS:
Overall Officials: Jimmi Elers, MD, Principal Investigator — Bispebjerg Hospital, Respiratory Research Unit
Locations (1):
- Bispebjerg Hospital, Respiratory Research Unit, København NV, Denmark